CLINICAL TRIAL: NCT04010474
Title: Comparison of Surgical APGAR Score and Modified Surgical APGAR Score in Predicting Possible Postoperative Complications in Major Surgery
Brief Title: Surgical APGAR Score and Modified Surgical APGAR Score
Status: Completed | Type: Observational
Sponsor: Namigar Turgut (Other)
Responsible Party: Sponsor-Investigator, Namigar Turgut, Prof.Dr, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: 09.05.2017 658
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Complication; Mortality; Modified; Surgical Apgar Score
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Modified Surgical APGAR Score — Four intraoperative factors
  1. Lowest heart rate (HR),
  2. Lowest mean arterial pressure (MAP)
  3. Estimated blood loss
  4. Operation time

SUMMARY:
In this study we aimed to define a new modified SAS is to predict the incidence of postoperative complication and mortality in major abdominal and orthopedic surgery. We also identify the effectivity of this modified scoring system composed of the duration of operation in addition to the three intraoperative parameters of SAS.

ELIGIBILITY:
Inclusion Criteria:

* Subject has major surgery
* More than 18 years

Exclusion Criteria:

* Pregnant
* Younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective major surgery (Abdominal and Orthopedic surgery) were included (n=308)
  After the operation modified SAS (mSAS) was calculated by adding the duration of the operation to data used in calculation of the SAS (Table 1.).
  Observed complications and related conditions were also noted.
  Table 1. Modified Surgical Apgar Score (mSAS)
  mSAS 0 1 2 3 4
  Estimated blood loss, ml >1000 601-1000 101-600 ≤100 -
  Lowest MAP*, mmHg <40 40-54 55-69 ≥70 -
  Lowest HR**, beats per min >85 76-85 66-75 56-65 ≤55
  Time -4 -3 -2 -1 0
  Duration of operation (hour) >8 7.01-8 5.01-7 3.01-5 0-3
  * MAP=Mean arterial pressure
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Surgical APGAR Score and Modified Surgical APGAR Score in Predicting Possible Postoperative Complications in Major Surgery | 01.06.2017 - 30.09.2017
  Operation time should be included as a simple, objective and practical indication of the SAS risk score in the major operations in our study including a single-center, prospective 308 case study, as it can be seen as an independent predictor of postoperative mortality and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Namigar Turgut, Prof.Dr, Study Director — University of Health Seciences, Okmeydani Training and Research Hospital
Locations (1):
- Namigar Turgut, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No